CLINICAL TRIAL: NCT01911143
Title: A Retrospective, Blinded Validation Study to Assess the Accuracy of a Host-response Based Diagnostics for Distinguishing Between Bacterial and Viral Etiologies in Pediatric Patients With an Acute Febrile Disease
Brief Title: A Retrospective, Blinded Validation of a Host-response Based Diagnostics
Acronym: PATHFINDER
Status: Completed | Type: Observational
Sponsor: MeMed Diagnostics Ltd. (Industry)
Collaborators: Bnai Zion Medical Center (Other Government); University Hospital, Geneva (Other)
Responsible Party: Sponsor
Other Study IDs: MM-1002-BV
Record Dates: First submitted 2013-07-15; First posted 2013-07-30 (Estimated); Last update posted 2016-03-08 (Estimated); Status verified 2016-03

CONDITIONS: Fever; Respiratory Tract Infections; Urinary Tract Infections; Gastroenteritis; Arthritis, Infectious
MeSH Terms: conditions — Fever; Respiratory Tract Infections; Urinary Tract Infections; Gastroenteritis; Arthritis, Infectious

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Biospecimen Retention: Samples Without DNA — Serum samples
Oversight: Data Monitoring Committee: No

SUMMARY:
This is a retrospective, blinded, external validation study of a novel in-vitro diagnostic (IVD) assay that will include samples that were previously collected from febrile pediatric patients. The investigated assay measures the levels of a few host-related, blood-based, bio-markers that will be integrated into a single score. Based on this score, each patient will be classified into one of three categories: (i) bacterial immune response, (ii) viral immune response, and (iii) marginal immune response. The assay prediction and the patient diagnosis will than be unveiled and compared to determine their level of concordance.

ELIGIBILITY:
Inclusion Criteria:

The infectious disease samples should also fulfill the following criteria:

* The patient had a peak temperature ≥38°C (AND)
* Symptoms initiated ≤ 7 days before sampling

The non-infectious disease control group will include:

* Patients with a non-infectious disease

Exclusion Criteria:

* Another infection episode during the last 3 weeks before sampling
* Congenital immune deficiency (CID)
* A proven or suspected HIV-1, HBV, HCV infection
* Active hematological malignancy
* Current treatment with immune-suppressive or immune-modulating
* Other illnesses that affect life expectancy and/or quality of life

Ages: 1 Month to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: The study population will include patients aged 1 month to 18 years of age that were sampled both during emergency department (ED) visit or during hospitalization stay and were diagnosed with an acute infectious disease or a non-infectious disease. All samples are expected to fall into one of the following categories:
  1. Patients with an acute bacterial infection
  2. Patients with an acute viral infection
  3. Patients with an acute mixed co-infection (bacterial and viral)
  4. Patients with a non-infectious disease (control group)
Sampling Method: Probability Sample
Enrollment: 600 (Actual)
Dates: Start 2013-09; Primary Completion 2015-08 (Actual); Study Completion 2015-08 (Actual)

PRIMARY OUTCOMES:
The sensitivity and specificity of the assay in differentiating between bacterial and viral etiology of patients with an acute febrile disease | 0-7 days after the initiation of symptoms
  We will evaluate the assay using the accuracy measures sensitivity and specificity of differentiating between bacterial and viral etiology of pediatric patients aged 1 month to 18 years with an acute febrile disease.

SECONDARY OUTCOMES:
The sensitivity and specificity of the assay in differentiating between infectious and non-infectious disease etiology. | 0-7 days after the initiation of symptoms
  We will evaluate the assay using the accuracy measures sensitivity and specificity of differentiating between infectious and non-infectious disease etiology in pediatric patients aged 1 month to 18 years.

CONTACTS AND LOCATIONS:
Overall Officials: Kfir Oved, Dr., Study Director — MeMed Diagnostics Ltd.
Locations (2):
- Israel (2):
  - Hillel Yaffe Medical Center, Hadera
  - Bnai Zion Medical Center, Haifa

IPD SHARING:
Plan to Share IPD: No